CLINICAL TRIAL: NCT01279603
Title: A Phase 1, Multi-center, Open-label, Dose-escalation, Safety, Pharmacodynamic and Pharmacokinetic Study of GO-203-2c Given Intravenously Daily X21 Repeated Every 28 Days in Patients With Advanced Solid Tumors Including Lymphomas
Brief Title: Study of GO-203-2C Given Intravenously in Patients With Advanced Solid Tumors Including Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genus Oncology, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO-2C-001
Record Dates: First submitted 2011-01-11; First posted 2011-01-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Solid Tumors
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

ARMS (1):
- GO-203-2c (Experimental)
  Interventions: Drug: GO-203-2c

INTERVENTIONS:
Drug: GO-203-2c — GO-203-2c Injection is a non-preserved, sterile, ready-to-use liquid dosage form provided in a glass vial with rubber closure and crimp seal. Injection will be added to the contents of an intravenous bag (of 0.9% NS, D5W or sterile water) to a final concentration of between 0.03 - 0.3 mg/ml (preferable in 100 mls or greater) and administered as a single agent intravenously over 60 minutes. A treatment cycle will consist of a daily IV dose administered for 21 consecutive days followed by a 7 day rest.

SUMMARY:
This clinical trial is about testing GO-203-2c, which is a newly discovered compound that binds to an oncoprotein (a cancer causing protein) called MUC1 (which is over-expressed in many cancers). By binding to MUC1, GO-203-2c eventually causes tumor cell death in laboratory studies.

This study is being done to:

* Test the safety of GO-203-2c and see what effects (good and bad) it has on you and your cancer
* Find the highest dose of GO-203-2c that can be given without causing bad side effects
* Examine how much GO-203-2c is in the blood at certain times after it is given and how quickly the body gets rid of it
* Observe whether there is any effect of GO-203-2c on the size and activity of cancer in your body

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumors or lymphomas
* Tumor progression observed after receiving standard/approved systemic chemotherapy and/or immunotherapy including monoclonal antibodies, or when there is no approved or effective therapy
* One or more measureable tumors by radiological evaluation
* Karnofsky performance ≥ 70%
* Life expectancy of ≥ 3 months
* Age ≥ 18 years
* Signed, written IRB-approved informed consent
* Negative pregnancy test (if female)
* Adequate liver function:
* Bilirubin less than or equal to 1.5 x upper limit of normal (ULN)
* AST (SGOT), ALT (SGPT) and Alkaline phosphatase less than or equal to 2.5 x ULN (if liver metastases are present, then less than or equal to 5 x ULN is allowed)
* Adequate renal function:
* Serum creatinine within normal limits, OR calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with serum creatinine above institutional ULN.
* Corrected serum calcium ≥ lower limit of the institutional normal range (LLN)
* Serum phosphorus level ≥ LLN
* Adequate hematologic function:
* Absolute Neutrophil Count ≥ 1500 cells/mm3
* Platelet count ≥ 100,000 (cells/mm3)
* Hemoglobin ≥ 9 g/dL
* Urinalysis:
* No clinically significant abnormalities
* Adequate coagulation function:
* PT ≤ 1.25 x ULN
* PTT ≤ 1.25 x ULN
* For men and women of child-producing potential, agreement to use effective contraceptive methods during the study

Exclusion Criteria:

* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG
* Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy
* Pregnant or nursing women. NOTE: Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately.
* Major surgery within 4 weeks prior to Day 1, or not fully recovered by Day 1
* Minor surgery within 2 weeks prior to Day 1, or not fully recovered by Day 1
* Treatment with radiation therapy within 4 weeks prior to Day 1.
* Received systemic chemotherapy or monoclonal antibody or other immunotherapy within 4 weeks prior to Day 1 (exceptions: 6 weeks for nitrosourea, mitomycin C, or any agent with a known treatment effect > 4 weeks' duration), or not fully recovered from any side effects from previous therapy by Day 1
* History of allergic reactions attributed to excipients or chemical products used in the final GO-203-2c drug formulation
* Known infection with HIV, hepatitis B, or hepatitis C.
* Subjects with risk factors for gastrointestinal perforation or pulmonary hemorrhage (e.g. unresected luminal intestinal cancers; abdominal carcinomatosis within 3 months before the first dose of study drug, abdominal fistula, acute diverticulitis, peptic ulcer disease, irritable bowel syndrome, Crohn's disease, pulmonary hemorrhage, hemoptysis, or tuberculosis)
* Currently receiving or having received treatment with any other investigational agent within 4 weeks prior to Day 1, or not fully recovered from toxicities of prior treatment by Day 1
* Serious and/or poorly controlled non-malignant disease (including but not limited to, ongoing or active infection, hydronephrosis, hypertension, diabetes, or other conditions) that could compromise protocol objectives in the opinion of the Investigator and/or the sponsor. Patients with such conditions should be discussed with the Medical Monitor prior to enrollment. All medical conditions must be NCI CTCAE Grade 1 or lower at baseline.
* Unwillingness or inability to comply with requirements of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 months
  To determine the maximum tolerated dose (MTD) and identify the dose limiting toxicities (DLT) of GO-203-2c - To establish the dose of GO-203-2c recommended for future phase II protocols

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - TGen Clinical Research Service, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Gorodetska I, Samusieva A, Lahuta T, Ponomarova O, Socha O, Kozeretska I. Exploring New Frontiers: Alternative Breast Cancer Treatments Through Glycocalyx Research. Breast J. 2025 May 22;2025:9952727. doi: 10.1155/tbj/9952727. eCollection 2025. PMID 40443562